CLINICAL TRIAL: NCT06190769
Title: Prevalence Of Musculoskeletal Disorders Among Monks And Nuns In Egypt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, MARIAN MAGDY, Marian Magdy Zaky Ebrahim, Cairo University
Other Study IDs: 012/004804
Record Dates: First submitted 2023-12-08; First posted 2024-01-05 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Musculoskeletal Disorders; Prevalence
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation study - cross-sectional survey.: sample size of monks will be 400 subjects of both genders (monks and nuns) randomly selected from different monasteries, Participants aged from 24 years old and above thought monastic years. As:
  * (1-3) years novice or probationary
  * (4-10) years of monasticism
  * more than 10 years of monasticism

SUMMARY:
1. Sample size will be 400.
2. Age starts from 24 years old and more.
3. Body mass index ( BMI ) between 18.5 to 24.9 kg/m2
4. Years of ordination

   * (1-3) years novice or probationary
   * (4-10) years of monasticism.
   * more than 10 years of monasticism.
5. Samples will be selected from several monasteries in Egypt.
6. All data collected by Arabic version of Nordic questionnaire.

DETAILED DESCRIPTION:
Study design: Observation study - cross-sectional survey.

Participants: sample size of monks will be 400 subjects of both genders (monks and nuns) randomly selected from different monasteries, Participants aged from 24 years old and above thought monastic years. As:

* (1-3) years novice or probationary
* (4-10) years of monasticism
* more than 10 years of monasticism

ELIGIBILITY:
Inclusion Criteria:

1. Both genders will include in study.
2. Monks and nuns work in different works administration.
3. Age starts from 24 years old and more.
4. Body mass index (BMI) between 18.5 to 24.9 kg/m2

Exclusion Criteria:

1. Monk or nun had musculoskeletal abnormalities due to causes (congenital or traumatic).
2. Monk or nun with previous operation involving locomotor system.
3. Outside body mass index range.

Min Age: 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Monks and Nuns
Study Population: both genders (monks and nuns) randomly selected from different monasteries
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2024-02-25 (Estimated); Study Completion 2024-03-03 (Estimated)

PRIMARY OUTCOMES:
correlation between the daily life of monks and musculoskeletal disorders by Nordic Musculoskeletal Questionnaire | 1 year
  Nordic Musculoskeletal Questionnaire explains that the daily life of monk affected on musculoskeletal disorders but not prevented him from his praying

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H EL Gendy, professor, Study Director — supervisor of research
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
nordic questionaire

REFERENCES:
- [Background] Vieira ER, Schneider P, Guidera C, Gadotti IC, Brunt D. Work-related musculoskeletal disorders among physical therapists: A systematic review. J Back Musculoskelet Rehabil. 2016 Aug 10;29(3):417-28. doi: 10.3233/BMR-150649. PMID 26577282

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/69/NCT06190769/SAP_000.pdf